CLINICAL TRIAL: NCT04861506
Title: Physician-initiated, Prospective, Multi-center, Observational Study: The Safety and Efficiency Result of Endovascular Treatment of Acute or Subacute Thromboembolic Occlusions of Lower Extremity.
Brief Title: The Safety and Efficiency of Endovascular Treatment of Acute or Subacute Thromboembolic Occlusions of Lower Extremity.
Status: Recruiting | Type: Observational
Sponsor: First People's Hospital of Hangzhou (Other)
Collaborators: RenJi Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Xuanwu Hospital, Beijing (Other); Qingdao Haici Hospital (Other); Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other); Second Affiliated Hospital of Suzhou University (Other); Chengdu University of Traditional Chinese Medicine (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Fangxin, Hospital director, Hangzhou Cancer Hospital
Other Study IDs: The Resolve Study
Record Dates: First submitted 2021-04-11; First posted 2021-04-27 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Thromboembolic Disease; Lower Extremity Problem; Endovascular Treatment; Safety Issues; Efficacy, Self
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- acute or subacute thromboembolic occlusions of lower extremity: The patients are confirmed with acute or subacute thromboembolic occlusions of lower extremity, and which are treated by endovascular therapy, through contralateral femoral artery approach, ipsilateral antegrade femoral artery approach or brachial artery approach. If the lesion is difficult to pass in antegrade approach, retrograde puncture at the distal artery of the lesion can be performed. Surgeons can choose treatment methods such as mechanical thrombectomy device (MTD) and/or pharmacomechanical thrombectomy (PMT）and/or percutaneous aspiration thrombectom (PAT) and/or CDT(catheter-directed thrombolysis) and/or percutaneous aspiration thrombectom (PAT) for thrombus removal according to the characteristics of the lesions and hospital conditions.
  Interventions: Procedure: endovascular treatment

INTERVENTIONS:
Procedure: endovascular treatment — All the patients are treated by endovascular therapy, through contralateral femoral artery approach, ipsilateral antegrade femoral artery approach or brachial artery approach. If the lesion is difficult to pass in antegrade approach, retrograde puncture at the distal artery of the lesion can be performed. Surgeons can choose treatment methods such as pharmacomechanical thrombectomy (PMT) and mechanical thrombectomy device (MTD) and/or pharmacomechanical thrombectomy (PMT）and/or percutaneous aspiration thrombectom (PAT) and/or CDT(catheter-directed thrombolysis) and/or percutaneous aspiration thrombectom (PAT) thrombolysis (CDT) for thrombus removal according to the characteristics of the lesions and hospital conditions.

SUMMARY:
Based on the development of new tools, including drug coated balloon, paclitaxel eluting stent, interwoven stents, debulking tools, More and more acute or subacute thromboembolic occlusions of lower extremity included stage IIb were treated with endovascular procedures. Most guidelines suggests only stage I and stage IIa lesions are suitable for endovascular treatments. Therefore, a well-designed real-world study that track the safety and clinical relevant outcomes, are required to determine the optimal therapies for patients with acute or subacute thromboembolic occlusions of lower extremity.

DETAILED DESCRIPTION:
According to the Trans-Atlantic Inter-Society Consensus (TASC) II guidelines, acute arterial occlusion which in stage IIb was recommended for thrombectomy. However, with the development of new tools, including drug coated balloon, paclitaxel eluting stent, interwoven stents, debulking tools, stage IIb patients and some subacute thromboembolic lesions were also effective in some retrospective studies.

Despite The shift of Endovascular-first strategy has been documented in recent literature. There still lack evidence to support either approach have a significant advantage over the thrombectomy. And stage IIb lesions and subacute lesions are often excluded in prospective clinical trials. Therefore, a well-designed real-world study that track the safety and clinical relevant outcomes, are required to determine the optimal therapies for patients with acute or subacute thromboembolic occlusions of lower extremity.

ELIGIBILITY:
Inclusion criteria

1. Patients aged 18 years or older.
2. Diagnosis of acute or subacute limb ischemia classified as Rutherford classification stage I to IIb.
3. Rutherford classification ranging from 3 to 5.
4. Successful guidewire passage through the lesion of the femoropopliteal artery lesion, followed by further endovascular treatment. There are no restrictions will be implemented on the methods used for guidewire passage through the target lesion. The presence of thrombus must be confirmed via angiography and/or DSA and must be associated with occlusions of the lower extremity or ISR.
5. Mechanical thrombectomy device (MTD) and/or pharmacomechanical thrombectomy (PMT) and/or percutaneous aspiration thrombectomy(PAT) and/or CDT (catheter-directed thrombolysis) performed for thrombus removal.
6. The lower extremity artery must have a healthy runoff of at least 10 cm above the ankle with at least one healthy dorsalis pedis artery, medial plantar artery, or lateral plantar artery connecting to the digital artery below the ankle.
7. Informed consent signed by patients.

Exclusion criteria

1. Acute or subacute limb ischemia patients with Rutherford classification stage III.
2. Patients diagnosed with thromboangiitis obliterans.
3. Patients requring open surgery or hybrid operation after contrast radiography.
4. Patients with a history of stroke, cerebral hemorrhage, gastrointestinal bleeding, myocardial infarction, or similar conditions in the past 3 months.
5. Patients with known allergies to heparin, low molecular weight heparin, or contrast agents.
6. Patients at high risk for bleeding.
7. Pregnant or lactating women.
8. Patients with other conditions that may complicate study participation or significantly reduce life expectancy (< 2 years), such as tumors, severe liver disease, and cardiac insufficiency.
9. Patients enrolled in other clinical studies within the past 3 months.
10. Patients unwilling or refusing to sign the informed consent form.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute or subacute thromboembolic occlusions of lower extremity who undergoing endovascular treatment.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Amputation-free survival | post-interventional 12months
  The amputation-free survival after endovascular surgery
Adverse events at post-interventional 1months | post-interventional 1 months
  the incidence of amputation, operation-related distal embolism, rethrombosis, acute renal failure and/or death.

SECONDARY OUTCOMES:
Technical success rate | Post operation up to 1 day
  Technical success rate
Clinical-driven Target lesion reintervention(CD-TLR) rate | post-interventional 12 months
  Clinical-driven Target lesion reintervention rate
Clinical-driven Target vascular reintervention(CD-TVR) rate | post-interventional 12 months
  Clinical-driven Target vascular reintervention rate
The total time used in the operation | Intraoperative
  The total time used in the operation
Primary patency(PP)of the lesions | post-interventional 12 months
  Primary patency(PP)of the lesions
Changes of quality of life assessed by VascuQol scale | post-interventional 12 months
  Changes of quality of life
Direct medical expenses (2-year cumulative hospitalization expenses and endovascular expenses related to target lesions) | 2 years
  Direct medical expenses

CONTACTS AND LOCATIONS:
Overall Officials: Meng Ye, Principal Investigator — RenJi Hospital; Ziheng Wu, Principal Investigator — First Affiliated Hospital of Zhejiang University; Lianrui Guo, Principal Investigator — Xuanwu Hospital, Beijing; Qiang Li, Principal Investigator — Qingdao Haici Hospital; Zibo Feng, Principal Investigator — Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology; Hongfei Sang, Principal Investigator — Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology; Chunshui He, Principal Investigator — Chengdu University of Traditional Chinese Medicine; Zhenyu Shi, Principal Investigator — Shanghai Zhongshan Hospital; Xupin Xie, Principal Investigator — First People's Hospital of Hangzhou; Jianyun Long, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Fan xin, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Long J, Wang L, Huang C, Xie X, Liu Y, Chen Y, Liu H, Ni Q, Yang S, Wu Z, Guo L, Feng Z, Li Q, He C, Sang H, Shi Z, Ye M, Fang X. Design of the RESOLVE study: a prospective, multicentre, observational, cohort study evaluating the safety and efficacy of endovascular treatment for acute or subacute thromboembolic occlusions of the lower extremity in China. BMJ Open. 2025 Oct 14;15(10):e103283. doi: 10.1136/bmjopen-2025-103283. PMID 41087108